CLINICAL TRIAL: NCT04021212
Title: Effects of Pituitary Adenoma Resection on Serum Lipid Level
Brief Title: Pituitary Adenoma and Serum Lipid
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Jia-jun Zhao, Principal Investigator, Shandong Provincial Hospital
Other Study IDs: 20190712
Record Dates: First submitted 2019-07-15; First posted 2019-07-16 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Pituitary Adenoma 1, Acth-Secreting
Keywords: Pituitary; Pituitary Adenoma; Serum Lipid Levels; Resection; Recurrence
MeSH Terms: conditions — Pituitary Diseases; Pituitary Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum，plasma, whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with pituitary adenomas resection: Patients suffers from pituitary adenomas and undergo transsphenoidal surgery for at least once

SUMMARY:
Pituitary adenomas are usually benign monoclonal neoplasms caused by a mixture of pituicyte alterations together with a changed endocrine and paracrine regulatory milieu. Thus, it can cause serious health problems such as abnormal target organ function, pain, disability and even death. In clinical practice, we found many patients with pituitary adenomas are usually accompanied by hyperlipidemia, which is the main cause of cardiovascular diseases. However, it has been unclear if there is an association between pituitary adenomas and serum lipid profile. In the present study, we aim to focus on the patients with pituitary adenomas and their lipid profile before and after operation including first occurrence and recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with pituitary adenomas
2. All adenomas were resected by transsphenoidal surgery and identified by histological diagnoses.

Exclusion Criteria:

1. Missing vital data, such as age, gender, serum lipid profile, pathology reports;
2. Complications or conditions that affect pituitary status and lipid metabolism, such as pregnancy, malignant adenomas or severe hepatic or renal dysfunction and
3. Use of any medication that affects the pituitary or lipid metabolism, including statins, fibrates, thyroid hormones, anti-thyroid drugs, iodine, amiodarone, alemtuzumab, lithium, tyrosine kinase inhibitors, interferon, estrogens, androgens,glucocorticoids, nonsteroidal anti-inflammatory drugs, antiepileptic drugs, rifampicin, furosemide, heparin or β-adrenoceptor blockers in the past 3 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with pituitary adenomas and underwent an endoscopic transsphenoidal approach at the Shandong Provincial Hospital affiliated with Shandong University. All adenomas were resected by transsphenoidal surgery and identified by histological diagnoses.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change in serum lipid levels | Measured at pre-operative and 6 months after operation

CONTACTS AND LOCATIONS:
Overall Officials: Jiajun Zhao, Study Chair — Shandong Provincial Hospital
Locations (1):
- Shandong Provincial Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided